CLINICAL TRIAL: NCT01302405
Title: A Phase Ia/Ib Clinical Trial of PRI-724 in Patients With Advanced Solid Tumors
Brief Title: Safety and Efficacy Study of PRI-724 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: closing due to low enrollment, no safety issues
Sponsor: Prism Pharma Co., Ltd. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRI-724-101
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2015-10

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumor; cancer; phase 1; pancreatic cancer; colon cancer; unresectable neoplastic disease; Progressive cancer; metastatic solid tumor
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Neoplasm Metastasis | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRI-724 (Experimental)
  Interventions: Drug: PRI-724

INTERVENTIONS:
Drug: PRI-724 — Dose escalation

SUMMARY:
PRI-724 is a new investigational drug being studied to treat subjects with cancer who have advanced solid tumors. PRI-724 is thought to work by blocking the Wnt signaling pathway that cancer cells need to grow and spread(metastasize).

Phase Ia: Patient cohorts with solid tumor malignancies will be treated with escalating doses (per cohort) of PRI-724 in order to identify the MTD of this single-agent regimen. PRI-724 dosing is to start at 40 mg/m2/day, CIV infusion over 24 hours × 7 days.

Phase Ib: This phase is to begin upon identification of the MTD in Phase 1a. Patient cohorts with CRC will be treated with escalating doses (per cohort) of PRI-724 administered in combination with a modified regimen of FOLFOX6 (mFOLFOX 6, standardized doses and schedule) in order to identify the MTD of this combined regimen. Up to 2 dose levels of PRI-724 are to be examined (640 and 905 mg/m2/day, CIV infusion over 24 hours × 7 days), with potential to evaluate a previously unexamined intermediate dose, if indicated, to more fully characterize tolerability. The MTD cohort (or maximum dose to be studied) will be expanded up to 12 patients.

DETAILED DESCRIPTION:
Primary Objectives

* Determine the MTD of PRI-724 when administered as a 7-day CIV intravenous infusion to patients with solid tumors (Phase Ia).
* Determine the MTD of PRI-724 when administered as a 7-day CIV infusion in combination with mFOLFOX6 in patients with colorectal carcinoma (Phase Ib).

Secondary Objectives

* Describe the dose-limiting toxicities (DLTs) and adverse event profile of PRI-724 when administered as a 7-day CIV infusion either alone in patients with solid tumors, or in combination with mFOLFOX6 in patients with colorectal carcinoma.
* Determine the pharmacokinetic (PK) profile of PRI-724 and C-82 when administered as a 7-day CIV infusion in these patient populations (In Phase 1b PK assessments will not be performed in expanded MTD cohort patients).
* Obtain preliminary assessment of anti-tumor activity as manifested by responses to treatment in these patient populations.
* Measure the mRNA expression of survivin by reverse transcriptase-polymerase chain reaction (RT-PCR), pre- and post-treatment with PRI-724:

  * In circulating tumor cells (CTC)
  * In tumor biopsy specimens from CRC patients (Phase Ib only) Also, evaluate whether survivin expression in CTC is consistent and reflective of expression in tumor specimens.
* Obtain preliminary assessments of potential associations of survivin that may be impacted by the pharmacodynamic (PD) properties of PRI-724 and clinical outcome, toxicity and PK parameters
* Assess the effects of Wnt inhibitor C-82 on the hair follicle neogenesis and the amount of collagen expression

Exploratory Objective

• Obtain matrix metalloproteinase-7 (MMP7) levels in serum via enzyme-linked immunosorbent assay (ELISA) testing

Study Design:

During the Phase Ia portion, an accelerated titration design, specifically, design 4A (no within-patient dose escalation) will be used, and will begin at the starting dose of 40 mg/m2/day. This involves an initial accelerated (double-step) dose escalation phase followed by a standard 3+3 design (single-step) dose escalation phase. In the initial accelerated phase, cohorts of one new patient will be treated per dose level and double-step dose escalations will be used. The accelerated phase will end when the first instance of DLT is observed during any cycle of treatment, or when a second patient experiences a moderate toxicity (MT) during any cycle. The cohort at the current dose level will be expanded and the standard 3+3 design phase (single-step) dose escalation will start for all subsequent cohorts.

In this study, the accelerated phase will end with Dose Level 9 (640 mg/m2/day), unless the toxicity criteria for terminating the accelerated phase are met earlier.

During the accelerated phase, decisions to escalate, expand, or de-escalate will be made when all patients at the current dose level have completed one cycle (2 weeks) of PRI-724, and have received at least 75% of the planned PRI-724 dose, or have experienced a MT or DLT.

During the standard 3+3 phase, decisions to escalate, expand, or de-escalate will be made when all patients at the current dose level have completed two cycles (4 weeks) of PRI-724 and have received at least 75% of the planned PRI-724 dose, or have experienced DLT.

During the Phase Ib portion, dose escalation in patients with CRC will begin at Level 9 of the doses evaluated during Phase Ia (640 mg/m2/day). Up to 2 dose levels will be evaluated (640 and 905mg/m2/day; potential to evaluate a previously unexamined intermediate dose, if indicated) using a standard 3+3 design (single-step dose escalation). Decisions to escalate, expand, or de-escalate will be made when all patients at the current dose level have completed two cycles (4 weeks) of PRI-724 plus mFOLFOX6 (i.e., 2 courses of PRI-724 and 2 courses of mFOLFOX6), and have received at least 75% of the planned PRI-724 dose, or have experienced a DLT.

In both Phase 1a and Phase 1b, the decision to escalate, expand, or de-escalate a cohort may be made by the Sponsor and the Investigator(s) in the absence of a defined DLT if it is determined that a dose level is impractical due to the frequency or nature of toxicities that do not meet DLT criteria. In such a case when a particular dose is deemed impractical, the next lower dose cohort may be expanded for further investigation. Once additional safety data are available, consideration may be given toward identifying the lower dose as the MTD or recommended Phase 2 dose.

Throughout the study, enrollment will be staggered between the first and second patient in each new cohort, to allow for one cycle (2 weeks) to elapse prior to enrolling the second patient into the cohort.

The following toxicities considered by the Investigator to be at least possibly related to study therapy (or study therapy plus chemotherapy) are defined as DLTs:

Non-Hematological DLTs:

* All Grade 3-4 non-hematologic toxicities that represent a 2 grade increase from baseline, excluding:

  * Untreated or inadequately treated nausea, vomiting and diarrhea
  * Alopecia
  * Grade 3 fatigue that returns to Grade 2 or lower within 7 days
* Grade 3 laboratory and/or metabolic abnormalities that do not return to Grade 2 or lower within 72 hours despite treatment
* QTcF > 500 msec OR an increase in QTc by 60 msec from baseline

Hematologic DLTs:

* Grade 4 neutropenia
* Grade 4 thrombocytopenia
* Neutropenic fever
* ≥ Grade 3 anemia unresponsive to supportive care including blood transfusion and/or erythropoietin therapy
* Grade 3 thrombocytopenia with clinically significant bleeding The DLT observation period, measured from the start of the infusion on the first day, is 2 weeks for the accelerated phase in the Phase Ia portion, and 4 weeks for the 3 + 3 phase in both the Phase Ia and Phase Ib portions of the trial.

Moderate toxicity (MT) is defined as any ≥ Grade 2 toxicity (except alopecia) that is considered by the Investigator to be at least possibly related to the study therapy and that does not qualify as a DLT.

During the Phase Ia portion, MTD is defined as the highest dose level tested in which no patient or only 1 patient experienced a DLT attributable to the study drug(s), when at least 6 patients were treated at that dose and are evaluable for toxicity. The MTD is one dose level below the maximally administered dose (MAD), which is the lowest dose level tested in which 2 or more patients experienced a DLT attributable to the study drug(s). In Phase Ia at least 6 patients will be treated at the MTD.

During the Phase Ib portion, the MTD is defined as the highest dose level tested in which no patient or only 1 patient experienced a DLT attributable to the study drug(s), when at least 6 patients were treated at that dose and are evaluable for toxicity, or when < 33.3% of patients experienced a DLT attributable to the study drug(s) when 7 to 12 patients were treated at that dose and are evaluable for toxicity. (This would allow for up to 2 DLTs when 7 to 9 patients have been enrolled in the expansion cohort or up to 3 DLTs when 10 to 12 patients have been enrolled in the expansion cohort.) The MTD is one dose level below the MAD which is the lowest dose tested in which> 1 patient in a 3- to 6-patient cohort, or > 33.3% of patients in an expanded 7- to 12-patient cohort, experienced a DLT attributable to the study drug(s). In Phase Ib at least 12 patients will be treated at the MTD.

There is potential for expansion of a lower dose cohort up to 12 patients if the initially identified and expanded MTD cohort is found to exceed tolerability.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfill all of the following criteria:

1. In the dose-escalation part of the study (Phase Ia), patients mu have histological or cytological evidence of solid tumor malignancy; in the tumor-specific, dose-escalation/MTD-expansion part of the study (Phase Ib), patients must have histological or cytological evidence of colorectal cancer.
2. Patients must have neoplastic disease that is metastatic or unresectable, that has recurred or progressed following standard therapy, not be candidates for standard therapy, or have a malignancy for which no standard therapy exists. In Phase Ib,patients must have colorectal cancer with tumor sites safely accessible for biopsy, and they must have measurable disease according to the response evaluation criteria in solid tumors (RECIST 1.1) criteria.
3. In Phase Ib patients must have received and either relapsed from or failed at least two but no more than three prior regimens of chemotherapy, and be eligible to receive third- or fourth-line therapy for their malignancy.
4. Patients must agree, as part of the informed consent, to provide blood samples for molecular correlative studies. In the Phase Ib cohorts, patients must agree to pre- and post-treatment biopsies of their malignant disease.
5. Patients must be > 18 years of age.
6. Patients must have a Karnofsky Performance Score of 70% - 100%.
7. Patients must have a life expectancy of at least 12 weeks.
8. Patients or their legal representatives must be able to comprehend and provide written informed consent.
9. Patients must have adequate bone marrow reserve as evidenced by:

   * White blood cell (WBC) count> 3,000/µL
   * Absolute neutrophil count (ANC) > 1,500/µL - Platelet count> 100,000/µL
10. Patients must have adequate renal function as evidenced by a serum creatinine value less than the upper limit of normal (< ULN) for the reference lab or creatinine clearance (CrCl) of > 60 mL/min (as calculated by Cockcroft-Gault formula).
11. Patients must have adequate hepatic function as evidenced by a serum bilirubin < 1.5 mg/dL and serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels < 3X the ULN for the reference lab (< 5X the ULN if there is evidence of hepatic involvement by malignant disease).
12. Patients must be recovered to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies. In Phase Ib patients must have no peripheral sensory neuropathy > Grade 1.
13. Women of childbearing potential (WOCBP) and male patients with WOCBP partner must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Postmenopausal is defined as:

    * Amenorrhea ≥12 consecutive months without another cause or
    * For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level> 35 mIU/mL.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of investigational product.

Exclusion Criteria:

Patients exhibiting any of the following will be excluded from the trial:

1. Infection requiring systemic antibiotics 72 hours prior to the first dose of PRI-724.
2. Known hypersensitivity to any of the components of PRI-724.
3. Women who are pregnant or lactating.
4. Untreated central nervous system (CNS) metastases; patients whose CNS metastases have been treated by surgery or radiotherapy, who are no longer on corticosteroids, and who are neurologically stable may be enrolled in the initial dose escalation portion of the trial (Phase Ia), but not in the Phase Ib portion of the trial.
5. Treatment with any investigational agent within a period of 28 days between the last dose of the investigational agent and the first dose of PRI-724.
6. QTcF intervals > 470 msec (females) or > 450 msec (males).
7. Active hepatitis B, hepatitis C.
8. New York Heart Association (NYHA) Class 3 or 4; myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months; or any other intercurrent medical condition that contra-indicates treatment with PRI-724 or places the patient at undue risk for treatment-related complications.
9. Any other condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
10. Patients with a current condition of osteopenia or osteoporosis via a Dual Energy X-ray Absorptiometry (DEXA) scan; patients with a history of either are allowed.
11. Patients on any dose of warfarin are excluded.
12. Given the potential interaction between C82, the metabolite of PRI-724, and CYP3A4 inhibitors, treating physicians should exercise caution and switch patients to equivalent drugs that are not potent CYP3A4 inhibitors when feasible. Medications which are sensitive substrates of CYP2C9 or CYP3A4 with a narrow therapeutic range should be used with caution.
13. In Phase 1b, patients with a history of poor FOLFOX tolerability as manifested by inability to tolerate standard therapeutic doses (i.e., at minimum patients must have tolerated an oxaliplatin dose of 85 mg/m2 and a 5FU dose of 2400 mg/m2).

Note: Patients are eligible for this trial if, during the previous FOLFOX administration, they underwent one dose reduction of oxaliplatin due to sensory neuropathy (provided the neuropathy has now resolved to Grade 1 or less), and/or one dose reduction of 5FU due to cumulative toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Maximum Therapeutic Dose, as defined by the highest dose identified in which ≤1/3 or ≤2/6 patients do not experience a dose limiting toxicity | Assessed at the completion of each patient enrollment cohort. Each patient monitoring duration is 28 days.
  Maximum Therapeutic Dose (MTD) will be the highest dose in which no dose limiting toxicity (DLT) is seen in a accelerated enrollment cohort (1 patient) and then subsequently a 3-6 patient cohort following a 3+3 study design. MTD may also be determined by evaluation of PK and PD results of patients.

SECONDARY OUTCOMES:
Maximum Therapeutic Dose of combined regimen, as defined by the highest dose identified in which ≤1/3 or ≤2/6 patients do not experience a dose limiting toxicity | Assessed at the completion of each patient enrollment cohort. Each patient monitoring duration is 28 days
  Maximum Therapeutic Dose (MTD) of the combined regimen will be the highest dose in which MTD is defined as the highest dose level tested in which no patient or only 1 patient experienced a DLT in a 3-6 patient cohort or less than 33.3% of 7 - 12 patients experienced a DLT in the 12-patient expansion cohort. MTD may also be determined by evaluation of PK and PD results of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic, Department of Oncology, Rochester, Minnesota